CLINICAL TRIAL: NCT00878072
Title: A Multicenter, Open-label, Single-arm Study to Evaluate the Safety and Pharmacokinetics of Famciclovir Single 1500 mg Dose in Adolescents With Recurrent Herpes Labialis
Brief Title: Safety and Pharmacokinetics of Famciclovir Single 1500 mg Dose in Adolescents With Recurrent Herpes Labialis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFAM810B2305
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Herpes Labialis
Keywords: Herpes labialis; cold sores; herpes simplex type 1
MeSH Terms: conditions — Herpes Labialis | interventions — Famciclovir

ARMS (1):
- Famciclovir (Experimental)
  Interventions: Drug: Famciclovir

INTERVENTIONS:
Drug: Famciclovir — Famciclovir 1500 mg (3 x 500 mg tablets) oral as a single dose.

SUMMARY:
This study will assess the safety, tolerability of a single 1500 mg dose of famciclovir in 50 adolescents with recurrent herpes labialis. Eight of the 50 adolescents will also participate in the pharmacokinetics (PK) assessment of famciclovir single 1500 mg dose

DETAILED DESCRIPTION:
Uncontrolled study

ELIGIBILITY:
Inclusion Criteria:

* Outpatient males or females 12 to <18 years of age
* General good health with a documented history typical for recurrent herpes labialis
* Prodromal symptoms or active lesions suggestive of a recurrent episode of herpes labialis (i.e. having had cold sores in the past) , with onset not exceeding 24 hours until the time of study drug administration

  * Adolescents participating in Pharmacokinetics (PK) part of the study may be enrolled without an active herpes labialis recurrence or with onset of signs/symptoms of a recurrent herpes labialis episode longer than 24 hours before study drug administration, All adolescents participating in the pharmacokinetics assessments must fast for at least 8 hours prior to Visit 1 and be willing to fast for an additional 2 hours after study drug administration

Exclusion Criteria:

* Use of other investigational drugs within 30 days of enrollment
* History of hypersensitivity to famciclovir or penciclovir
* Inability to swallow tablets
* Body weight less than 40 Killograms (kg)
* History of malabsorption, unless a condition like celiac disease is stable and well controlled, previous gastrointestinal surgery or radiation therapy that could affect drug absorption or metabolism, or any condition that could interfere with drug absorption, distribution, metabolism, or excretion
* Known renal insufficiency (calculated creatinine clearance <60 [Milliliters/Minutes] mL/min)
* Known severe hepatic impairment (Child-Pugh Class C)
* Significant skin disease such as atopic dermatitis or eczema that would interfere with assessment of oral/labial lesions
* Known to be immunocompromised or are receiving systemic or using topical immunosuppressive agents (including corticosteroids, tacrolimus and picrolimus) within 30 days of enrollment
* Concomitant use of probenecid
* Pregnant or nursing (lactating) females
* Females of child-bearing potential, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2009-03-25; Primary Completion 2010-06-02 (Actual); Study Completion 2010-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Women's Health Care at Frost Street, San Diego, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - Clayton Medical Research, St Louis, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Westover Heights Clinic, Portland, Oregon
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - R/D Clinical Research, Inc, Lake Jackson, Texas
  - R/D Clinical Research, Lake Jackson, Texas

REFERENCES:
- [Derived] Block SL, Yogev R, Waldmeier F, Hamed K. Safety and pharmacokinetics of a single 1500-mg dose of famciclovir in adolescents with recurrent herpes labialis. Pediatr Infect Dis J. 2011 Jun;30(6):525-8. doi: 10.1097/INF.0b013e3182067cee. PMID 21178655
- See also: NovartisClinicalTrials.com: pre-screening for this trial, view of a list of trials and participating study centers — http://www.adolescentcoldsoresstudy.com
- See also: Adolescent Cold Sores Clinical Trial — http://www.novartisclinicaltrials.com/webapp/portals/AdolescentColdSoresStudy/page.do

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 centers in United States.
Groups:
- Famciclovir: Participants received single oral doses of three 500 milligrams (mg) Famciclovir tablets on Day 1.
Period: Overall Study
Arm/Group | Famciclovir
Started | 53
Completed | 51
Not Completed | 2
Not completed — Withdrew consent | 2

BASELINE CHARACTERISTICS:
Population: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Arm/Group | Famciclovir
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reported Adverse Events (AEs), Serious Adverse Events (SAEs)
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: From Start of the Study up to Day 36
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Famciclovir (Participants Aged 12 to Less Than [<] 15 Years): Participants aged 12 to <15 years received single oral doses of three 500 milligrams (mg) Famciclovir tablets on Day 1.
- Famciclovir (Participants Aged 15 to Less Than [<] 18 Years): Participants aged 15 to <18 years received single oral doses of three 500 milligrams (mg) Famciclovir tablets on Day 1.
Arm/Group | Famciclovir (Participants Aged 12 to Less Than [<] 15 Years) | Famciclovir (Participants Aged 15 to Less Than [<] 18 Years)
Number analyzed (Participants) | 28 | 25
Participants
  Adverse Events | 6 | 6
  Serious Adverse Events | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Participants with laboratory values outside the defined normal range were graded as clinically significant laboratory abnormalities. Laboratory values were assessed according to the National Cancer Institute- Common terminology criteria for Adverse Events (NCI-CTCAE). Hematology, Urinalysis and clinical chemistry were reported .
Time Frame: From Start of the Study up to Day 36
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Famciclovir (Participants Aged 12 to Less Than [<] 15 Years) | Famciclovir (Participants Aged 15 to Less Than [<] 18 Years)
Number analyzed (Participants) | 28 | 25
Participants
  Hematology | 0 | 0
  Clinical chemistry | 0 | 0
  Urinalysis | 0 | 0

3. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Penciclovir (Active Metabolite From Famciclovir) and 6-deoxypenciclovir (First Intermediate Metabolite From Famciclovir)
Description: Tmax was defined as the time to reach maximum plasma concentration. Penciclovir (active metabolite from famciclovir) and 6-deoxypenciclovir (first intermediate metabolite from famciclovir) were determined by using a validated liquid chromatography/tandem mass spectrometry (LC/MS/MS) method. The limit of quantification was 0.15 microgram (µg)/milliliter (mL) for both compounds. Calculations were done in WinNonlin 5.0.1, using non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6 and 10 hours Post-dose
Population: The analysis was performed in PK (Pharmacokinetics) analysis set (PAS) population, defined as all participants who participated in the PK assessment part and who did not miss more than one PK blood sampling. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Median (Full Range); unit: Hours
Groups:
- Penciclovir (Participants Aged 12 to Less Than [<] 18 Years); 6-Deoxy Penciclovir (Participants Aged 12 to Less Than [<] 18 Years): Participants aged 12 to <18 years received single oral doses of three 500 milligrams (mg) Famciclovir tablets.
Arm/Group | Penciclovir (Participants Aged 12 to Less Than [<] 18 Years) | 6-Deoxy Penciclovir (Participants Aged 12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 8 | 8
Hours | 1 [0.83 to 3.00] | 1 [0.5 to 2.0]

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Penciclovir (Active Metabolite From Famciclovir) and 6-deoxypenciclovir (First Intermediate Metabolite From Famciclovir)
Description: Cmax was defined as the maximum observed plasma concentration. Penciclovir (active metabolite from famciclovir) and 6-deoxypenciclovir (first intermediate metabolite from famciclovir) were determined by using LC/MS/MS method. The limit of quantification was 0.15 µg/mL for both compounds. Calculations were done in WinNonlin 5.0.1, using non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6 and 10 hours Post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microgram (µg)/milliliter(mL)
Arm/Group | Penciclovir (Participants Aged 12 to Less Than [<] 18 Years) | 6-Deoxy Penciclovir (Participants Aged 12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 8 | 8
Microgram (µg)/milliliter(mL) | 9.37 (2.68) | 3.32 (2.36)

5. Secondary Outcome: Area Under the Plasma Concentration of Penciclovir (Active Metabolite From Famciclovir) and 6-deoxypenciclovir (First Intermediate Metabolite From Famciclovir)
Description: AUC 0-tlast was defined as the area under the plasma concentration-time curve from time zero up to the last quantifiable concentration (Clast) calculated by the linear trapezoidal rule. Penciclovir (active metabolite from famciclovir) and 6-deoxypenciclovir (first intermediate metabolite from famciclovir) were determined by using LC/MS/MS method. The limit of quantification was 0.15 µg/mL for both compounds. Calculations were done in WinNonlin 5.0.1, using non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6 and 10 hours Post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microgram(µg)/Milliliter(mL)*Hour(h)
Arm/Group | Penciclovir (Participants Aged 12 to Less Than [<] 18 Years) | 6-Deoxy Penciclovir (Participants Aged 12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 8 | 8
Microgram(µg)/Milliliter(mL)*Hour(h) | 30.80 (5.52) | 5.42 (3.58)

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC 0-infinity) of Penciclovir (Active Metabolite From Famciclovir) and 6-deoxypenciclovir (First Intermediate Metabolite From Famciclovir)
Description: AUC 0-infinity was defined as the area under the plasma concentration time curve from time zero to infinity = AUC 0-tlast + C last /λ z, where λz is the apparent elimination rate constant estimated by linear regression analysis of the terminal portion of the log-linear plasma concentration-time curve. Penciclovir (active metabolite from famciclovir) and 6-deoxypenciclovir (first intermediate metabolite from famciclovir) were determined by using LC/MS/MS method. The limit of quantification was 0.15 µg/mL for both compounds. Calculations were done in WinNonlin 5.0.1, using non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6 and 10 hours Post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microgram(µg)/Milliliter(mL)*Hour(h)
Arm/Group | Penciclovir (Participants Aged 12 to Less Than [<] 18 Years) | 6-Deoxy Penciclovir (Participants Aged 12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 8 | 6
Microgram(µg)/Milliliter(mL)*Hour(h) | 31.76 (5.53) | 6.61 (3.89)

7. Secondary Outcome: Apparent Terminal Elimination Half-Life (T½) of Penciclovir (Active Metabolite From Famciclovir) and 6-deoxypenciclovir (First Intermediate Metabolite From Famciclovir)
Description: T½ was defined as the apparent terminal elimination half-life= ln 2/ λz. Penciclovir (active metabolite from famciclovir) and 6-deoxypenciclovir (first intermediate metabolite from famciclovir) were determined by using LC/MS/MS method. The limit of quantification was 0.15 µg/mL For both compounds. Calculations were done in WinNonlin 5.0.1, using non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6 and 10 hours Post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Penciclovir (Participants Aged 12 to Less Than [<] 18 Years) | 6-Deoxy Penciclovir (Participants Aged 12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 8 | 6
Hours | 1.81 (0.22) | 0.78 (0.21)

8. Secondary Outcome: Apparent Oral Clearance of Penciclovir From Plasma (CL/F) of Penciclovir (Active Metabolite From Famciclovir)
Description: CL/F was defined as the apparent oral clearance of penciclovir from plasma = dose of famciclovir*0.7884/AUC 0-inf, where 0.7884 is the ratio of the molecular weight of penciclovir (253.3 g/mol) to famciclovir (321.3 g/mol). F is the bioavailability of penciclovir after oral administration of famciclovir. Penciclovir (active metabolite from famciclovir) and 6-deoxypenciclovir (first intermediate metabolite from famciclovir) were determined by using LC/MS/MS method. The limit of quantification was 0.15 µg/mL for both compounds. Calculations were done in WinNonlin 5.0.1, using non-compartmental methods.
Time Frame: Pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6 and 10 hours Post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Litres(L)/Hour(h)
Arm/Group | Penciclovir (Participants Aged 12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 8
Litres(L)/Hour(h) | 38.2 (6.1)

ADVERSE EVENTS:
Time Frame: From Start of the Study up to Day 36.
Arm/Group | Famciclovir (Participants Aged 12 to Less Than [<] 15 Years) | Famciclovir (Participants Aged 15 to Less Than [<] 18 Years) | Famciclovir
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/25 | 0/53
Other Adverse Events (participants affected / at risk) | 6/28 | 6/25 | 12/53
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Famciclovir (Participants Aged 12 to Less Than [<] 15 Years) (N=28) | Famciclovir (Participants Aged 15 to Less Than [<] 18 Years) (N=25) | Famciclovir (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 3
Headache (Nervous system disorders) | 1 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes